CLINICAL TRIAL: NCT00982501
Title: Investigation of Safety of WS®1442 in Slightly Overweight Subjects With Pilot Assessment of Pharmacodynamic Effects of WS®1442 on Endothelial Function
Brief Title: WS®1442 in Slightly Overweight Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Willmar Schwabe GmbH & Co. KG (Industry)
Responsible Party: Professor Josef Niebauer, M.D., Ph.D., Universitaetsinstitut fuer praeventive und rehabilitative Sportmedizin der Paracelsus Medizinischen Privatuniversitaet, Institut fuer Sportmedizin des Landes Salzburg, Lindhofstr. 20, 5020 Salzburg, Austria
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 501004.01.103
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Overweight
Keywords: (BMI 25-29,9 kg/m2)
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- WS® 1442 900 mg (Experimental)
  Interventions: Drug: WS® 1442 900 mg/d
- WS® 1442 1800 mg (Experimental)
  Interventions: Drug: WS® 1442 1800 mg/d
- Nordic walking training 2x30 min (Active Comparator)
  Interventions: Behavioral: Nordic walking training 2 x 30 min/week
- Nordic walking training 4x45 min (Active Comparator)
  Interventions: Behavioral: Nordic walking training 4x45 min/week

INTERVENTIONS:
Drug: WS® 1442 900 mg/d
  Arms: WS® 1442 900 mg
Drug: WS® 1442 1800 mg/d
  Arms: WS® 1442 1800 mg
Behavioral: Nordic walking training 2 x 30 min/week
  Arms: Nordic walking training 2x30 min
Behavioral: Nordic walking training 4x45 min/week
  Arms: Nordic walking training 4x45 min

SUMMARY:
The purpose of this study is to test:

1. Safety of 900 mg or 1800 mg of WS® 1442 per day in overweight subjects (BMI 25 to 29,9 kg/m²)
2. Pharmacodynamic effect of WS® 1442 on endothelial function versus nordic walking training in overweight subjects

DETAILED DESCRIPTION:
60 overweight subjects with a BMI of 25 to 29,9 kg/m2 are to be included. The safety of 900 mg/1800 mg per day WS® 1442 is determined by adverse events, laboratory parameters, vital signs as well as by a treadmill test at the beginning and the end of the study. Endothelial function measured before and after two different training modalities is compared to that measured before and after intake of two different doses of WS® 1442.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* male and female subjects aged 45-75 years
* untrained
* BMI between 25 and 29,9 kg/m²
* resting blood pressure in sitting position ≤ 140/90 mmHg
* inconspicuous ergometry

Exclusion Criteria:

* pregnancy or breastfeeding
* any other current medication
* intake of other hawthorn preparation or dietary supplements with possible influence on the interpretation of study results
* any known diseases
* alcohol or drug abuse/addiction
* nicotine abuse
* any known hypersensitivity to any of the ingredients of the investigated drug
* inability or inadequate ability to write or speak German
* not-postmenopausal women: positive pregnancy test or unsafe contraception
* any urinary test finding requiring diagnostic assessment or treatment
* deformation of the 2nd to 5th finger of both hands preventing an adequate measurement of endothelial function

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 weeks
Lab parameters | 12 weeks
Vital signs | 12 weeks
Treadmill test including lactate measurement | 12 weeks

SECONDARY OUTCOMES:
Endothelial function | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Josef Niebauer, M.D., Ph.D., Principal Investigator — University Institute of Sports Medicine, Prevention and Rehabilitation
Locations (1):
- University Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University Salzburg, Salzburg, Austria